CLINICAL TRIAL: NCT04293549
Title: In Vivo Evaluation of Corneal Nerves and Epithelial Healing After Treatment With Nerve Growth Factor for Neurotrophic Keratopathy
Brief Title: An 8-week Follow-up to Evaluate the Renewal of Corneal Nerves Structure and Function in Patients With Neurotrophic Keratopathy Treated With Recombinant Human Nerve Growth Factor (rhNGF) Eyedrops
Status: Completed | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Leonardo Mastropasqua, Study Director, Professor, G. d'Annunzio University
Other Study IDs: UChieti01
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Neurotrophic Keratopathy
MeSH Terms: interventions — cenegermin; Ophthalmic Solutions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- rhNGF group: Therapeutic contact lens use was discontinued during the duration of the study. Patients underwent clinical examination with corneal fluorescein staining, Schirmer I tear test, assessment of corneal sensitivity with Cochet-Bonnet aesthesiometer and morphological examination of the nerves by In Vivo Confocal Microscopy (IVCM) at baseline and after 4 and 8 weeks of treatment. Changes in the corneal epithelium and stroma were evaluated by slit lamp biomicroscopy and photo documentation of the cornea after fluorescein staining.
  Interventions: Drug: Cenegermin, recombinant human Nerve Growth Factor (rhNGF) eyedrops
- control comparator group: control comparator group was matched for age and gender and underwent assessment of corneal sensitivity with Cochet-Bonnet aesthesiometer and morphological examination of the nerves by In Vivo Confocal Microscopy (IVCM) at baseline.

INTERVENTIONS:
Drug: Cenegermin, recombinant human Nerve Growth Factor (rhNGF) eyedrops — rhNGF 20µg/ml (Cenegermin) eyedrops, 1 drop every 2 hours (6 times a day) for 8 weeks.
  Patients underwent clinical examination with corneal fluorescein staining, Schirmer I tear test, assessment of corneal sensitivity with Cochet-Bonnet aesthesiometer and morphological examination of the nerves by In Vivo Confocal Microscopy (IVCM) at baseline and after 4 and 8 weeks of treatment
  Other Names: Oxervate
  Groups: rhNGF group

SUMMARY:
A prospective, longitudinal, cross-sectional, observational Study with a 8-week Follow-up to evaluate the renewal of corneal nerves structure and function in patients with Neurotrophic Keratopathy treated with recombinant human Nerve Growth Factor (rhNGF) eyedrops.

DETAILED DESCRIPTION:
This Study shows that topical treatment with Recombinant Nerve Growth Factor (rhNGF) improved corneal sensitivity and increased sub-basal nerves density, promoting corneal healing of persistent epithelial defects and corneal ulcers in patients with stage 2 and 3 NK

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented moderate or severe neurotrophic keratopathy based on a recent new classification of NK, refractory to conventional non surgical treatments. The diagnosis was made on medical and ophthalmological history, slit lamp examination, aesthesiometry, in vivo confocal microscopy.
* Decreased corneal sensitivity on the area of corneal defect and on superior, inferior, nasal and temporal quadrants (≤ 4 cm using the Cochet-Bonnet aesthesiometer)
* Patients who satisfy all Informed Consent requirements. The patient and/or his/her legal representative must read, sign and date the Informed Consent document before any study-related procedures are performed
* Patients with ability to understand and perform the treatment.

Exclusion Criteria:

* active infective keratitis or inflammation not related to NK in the affected eye.
* presence of corneal dystrophies.
* presence of glaucoma.
* Any other ocular disease requiring topical ocular treatment during the course of the study treatment period.
* History of any ocular surgery (including laser or refractive surgical procedures) within the three months before study enrolment. (An exception to the preceding statement will be allowed if the ocular surgery is considered to be the cause of the stage 2 or 3 NK).
* patients with known hypersensitivity to one of the components of the study or procedural medications (e.g. anaesthetic drops, fluorescein).
* Females currently pregnant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 18 patients (9 males and 9 females) were recruited from the Ocular Surface Service of G. d'Annunzio University of Chieti- Pescara and from the Division of Clinical Neuroscience, Department of Ophthalmology, University of Nottingham.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Changes of sub-basal nerve density, diameter and number of nerve branches | 8 weeks
  evaluated by In Vivo Confocal Microscopy (IVCM). Confocal microscopic scanning was focused on central cornea and superior, inferior, nasal and temporal quadrants; for each zone, 5 frames at the level of the epithelium and basal lamina were obtained. Corneal sub-basal nerve morphology and density was traced using NeuronJ, plug-in of ImageJ. Nerve regeneration rate was calculated.

SECONDARY OUTCOMES:
Changes in Corneal Sensitivity | 8 weeks
  measured by the Cochet-Bonnet aesthesiometer at 4 and 8 weeks after start of the treatment. Corneal sensitivity is measured in each patient in cm. the filament was applied on the area of corneal defect and on superior, inferior, nasal and temporal quadrants.
Changes of persistent epithelial defect and corneal ulcers | 8 weeks
  determined by corneal fluorescein staining at 4, 8 weeks as defined by the central reading center on clinical pictures

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Mastropasqua, Professor, Principal Investigator — Ophtalmology Clinic, G. d'Annunzio University
Locations (1):
- Ophtalmology Clinic, G.d'Annunzio University, Chieti, Italy